CLINICAL TRIAL: NCT05529212
Title: Cardiopulmonary Bypass Ischemia/Reperfusion Injury and Postoperative Multiple Organ Dysfunction in Elder Patients
Brief Title: Cardiac Surgery and Postoperative Organ Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Second Affiliated Hospital of Third Military Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Organ Dysfunction during CPB
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood and tissue samples be collected for biochemical testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ischemic reperfusion injury — ischemic reperfusion injury is a pathological process in which the ischemic myocardium is restored to normal perfusion, but the tissue damage is progressively aggravated when the coronary artery supply is completely blocked after cardiopulmonary bypass surgery and then recanalised at a certain time.

SUMMARY:
The aim of the study is to identify the correlation between ischaemia reperfusion injury and postoperative multiorgan damage during cardiopulmonary cardiac surgery; and to investigate biomarkers that can predict postoperative organ damage in cardiac surgery.

DETAILED DESCRIPTION:
This study proposes to observe multi-organ functional impairment of the heart, kidney and brain after extracorporeal circulation in a prospective study of clinical patients; to obtain markers with diagnostic and predictive efficacy by collecting pre and postoperative serum and heart and ear tissue samples from patients with postoperative organ functional impairment, performing combined proteomic and metabolomic analyses, and by analysing them with detailed postoperative clinical prognostic data using machine learning algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50 years; patients requiring mitral valve replacement surgery or mitral valve plus aortic valve replacement under cardiopulmonary bypass
2. Agreed to participate in this study, and signed the informed consent form.

Exclusion Criteria:

1. History of neurological disease (stroke, reversible ischemic hypoxia, transient ischemic attack, or Neurodegeneration) ;
2. Patients with severe preoperative renal insufficiency (serum creatinine > 442 μmol/L or need renal replacement therapy) ,
3. liver dysfunction (Child-Pugh grade C)
4. myocardial infarction within 4 weeks
5. ASA grade ≥ V

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were screened from the outpatient clinics of the Second Hospital of the Army Medical University who were proposed for mitral valve replacement or mitral valve combined with aortic valve replacement, agreed to participate in this study, and signed an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-16 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative cardiac injury | from the ending of surgery to 7 days after surgery
  troponin I will be tested before and after surgery
incidence of postoperative acute kidney injury | from the ending of surgery to 7 days after surgery
  renal function will be tested before and after surgery
incidence of postoperative brain injury | from the ending of surgery to 7 days after surgery
  deliriumwill be tested before and after surgery

SECONDARY OUTCOMES:
Incidence of postoperative arrhythmia events | from the ending of surgery to 72 hours after surgery
  postoperative arrhythmia events are recorded according to follow-up visits after surgery

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Chongqing Medical University, the second affiliated hospital
Locations (1):
- The second affiliated hospital of Chongqing medical university, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years